CLINICAL TRIAL: NCT03128125
Title: Study of Gesture and Executive Functions in Children With High Intellectual Potential
Acronym: MOHPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MOHPI (RB 16.145)
Record Dates: First submitted 2017-03-22; First posted 2017-04-25 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: High Intellectual Potential; Children
MeSH Terms: interventions — Restraint, Physical; Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: Case-control study, monocentric.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intellectual potential (Experimental): Participation in the study involves the conduct of a clinical examination in neurology, the collection of anamnestic elements and a neuropsychological examination in children with high intellectual potential.
  Interventions: Other: clinical examination in neurology; Other: neuropsychological examination; Other: anamnestic elements
- Control (Other): Participation in the study involves the conduct of a clinical examination in neurology, the collection of anamnestic elements and a neuropsychological examination in control children with no particularities.
  Interventions: Other: clinical examination in neurology; Other: neuropsychological examination; Other: anamnestic elements

INTERVENTIONS:
Other: clinical examination in neurology — This examination is based on the movement of the child in a standing position (forward and backward on a straight line, jumping on a foot ...), seated (visual continuation ...) and elongated (tone, patellar and achillian reflexes, superficial sensitivity ...) . This makes it possible to evaluate all the neurological systems.
Other: neuropsychological examination — This examination is based on the use of standardized psychometric tools and validated with children, usually used in clinical practice.
Other: anamnestic elements — Several elements will be collected during the clinical interview to inform the history of the child's development, such as neonatal data (term of pregnancy, APGAR score ...), age of appearance of the first words , seating, walking, possible care, level of education ans level of education of the parents.

SUMMARY:
The main objective of this study is to determine whether children with high intellectual potential have gestural and / or executive difficulties compared to control children.

ELIGIBILITY:
Inclusion Criteria:

All participants :

* Informed consent of the child and both parents obtained
* Affiliated to Social Security
* Participants must be between 6 and 16 years of age.

Child with high intellectual potential :

* Score ≥ 130 on an intellectual efficiency scale administered by a psychologist

Control child :

* They will have to be intellectually efficient in the standard. To ensure this, the two sub-tests of the Intellectual Efficiency Scale (WISC-V) most closely correlated with intelligence (Vocabulary and Matrices) will be administered to them. Thus, the child must meet one of the following criteria in order to be included:
* Have two standard notes between -1 and +1 DS (between 7 and 13);
* Have one of its two notes between -1 and + 1DS (between 7 and 13) and the other between -2DS and <+ 2DS (between 5 and 15).

Exclusion Criteria:

All participants :

* Neurological history (epilepsy, cranial trauma, prematurity ...)
* Psychiatric history (Autistic Spectrum Disorder ...),
* Known genetic disease,
* Motor deficiency (eg hemiplegia),
* Elementary sensory disorder (auditory and visual) or insufficient command of French, limiting the understanding and participation in the study likely to impact the results to the protocol.
* Gnosic visual or linguistic deficiency.
* Sensory disorder
* Psychotropic Intake

Control child :

* High intellectual potential
* Known or suspected learning disability (no dyslexia-dysorthography, dysphasia, dyspraxia, dyscalculia).

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Neuropsychological assessment | 1 day
  Determine whether children with high intellectual potential have gestural and / or executive difficulties compared to control children with WISC-V scale (Wechsler).
Neurological assessments | 1 day
  Dysfunction (yes/no) for children with high intellectual potential compared to control children.
Neuropsychological assessment | 1 day
  Determine whether children with high intellectual potential have gestural and / or executive difficulties compared to control children. With Purdue Pegboard test.
Neuropsychological assessment | 1 day
  Determine whether children with high intellectual potential have gestural and / or executive difficulties compared to control children. With subtest Fluence Verbale (NEPSY-II)
Neuropsychological assessment | 1 day
  Determine whether children with high intellectual potential have gestural and / or executive difficulties compared to control children. With subtest of motricity (NEPSY-II)
Neuropsychological assessment | 1 day
  Determine whether children with high intellectual potential have gestural and / or executive difficulties compared to control children. With Rey test
Neuropsychological assessment | 1 day
  Determine whether children with high intellectual potential have gestural and / or executive difficulties compared to control children. With writing test (BHK)
Neuropsychological assessment | 1 day
  Determine whether children with high intellectual potential have gestural and / or executive difficulties compared to control children. With New card sorting test
Neuropsychological assessment | 1 day
  Determine whether children with high intellectual potential have gestural and / or executive difficulties compared to control children. With comportemental scale (BRIEF)
Neuropsychological assessment | 1 day
  Determine whether children with high intellectual potential have gestural and / or executive difficulties compared to control children. With M-ABC-II questionary

CONTACTS AND LOCATIONS:
Overall Officials: Sylviane PEUDENIER, Principal Investigator — CHRU Brest
Locations (1):
- University Hospital, Brest, France